CLINICAL TRIAL: NCT01598662
Title: Safety and Expulsion of Delayed Versus Immediate Postpartum Intrauterine Device Placement: A Randomized, Controlled Trial
Brief Title: Safety and Expulsion of Delayed Versus Immediate Postpartum Intrauterine Device Placement
Acronym: IUD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to secure funding
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Mary Elaine Stauble, Assistant Professor, University of Louisville School of Medicine, Department of Obstetrics, Gynecology & Women's Health, Generalist Division, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IUD Study B090743
Record Dates: First submitted 2012-04-13; First posted 2012-05-15 (Estimated); Results first posted 2018-07-26 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-08

CONDITIONS: Contraception
Keywords: IUD placement; contraception; postpartum; intrauterine device; expulsion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1: IUD insertion 6 Weeks after delivery (Active Comparator): Device:Levonorgestrel-releasing intrauterine device marketed as Mirena.
  Subjects randomized to interval placement will have their IUD placed in the office at six weeks postpartum or later. They must return for one visit within a month for a "string check".
  Interventions: Device: Mirena (levonorgestrel-releasing intrauterine system)
- 2: Immediate Post-placental insertion (Experimental): Device: Levonorgestrel-releasing intrauterine device marketed as Mirena
  Subjects randomized to immediate post-placental placement within 10 minutes of delivery will have an IUD placed manually under sterile technique and with ultrasound guidance. An ultrasound will be performed within two days postpartum to verify proper placement and again at approximately six weeks postpartum.
  Interventions: Device: Mirena (levonorgestrel-releasing intrauterine system)

INTERVENTIONS:
Device: Mirena (levonorgestrel-releasing intrauterine system) — The Mirena IUD is a levonorgestrel-releasing IUD which contains 52 mg levonorgestrel total and releases 20 mcg of hormone daily.
  Other Names: Mirena IUD

SUMMARY:
This is randomized controlled trial designed for pregnant women who deliver vaginally at the University of Louisville Hospital and desire to have an intrauterine device (IUD) inserted for postpartum contraception. After informed consent is obtained, eligible study participants will be randomized to receive the Mirena® IUD at the 6 week postpartum visit or within 10 minutes of delivery of the placenta following a normal vaginal delivery. The investigators seek to determine the expulsion rate and complication rate in subjects with IUD immediately after placental delivery compared to insertion at six weeks postpartum or later. The investigators hypothesize that immediate placement safe and has an acceptably low expulsion rate to merit earlier placement in the indigent population.

DETAILED DESCRIPTION:
Unintended pregnancy occurs in nearly half of all pregnancies in the United States. There are many barriers to implementation of long-term reversible contraception in the immediate postpartum period. In our indigent population, a survey of patients showed that nearly 60% of patients who chose an IUD while admitted postpartum never returned for placement, placing them at risk for early repeat pregnancy.

The intrauterine device is a safe and effective form of long-term reversible contraception when placed at 6 weeks postpartum or later with pregnancy rates of only 0.1%. The commercially available Mirena IUD contains levonorgestrel which is released slowly over five years, providing safe, reversible contraception and making menstrual flow much lighter.

This randomized controlled trial will compare traditional placement at 6 weeks or more postpartum versus immediate post-placental placement.

The investigators hypothesize that the expulsion rate of IUDs placed immediately postpartum will be acceptably low in an indigent population to still be cost effective. Studies from the world literature in Egypt and Mexico where IUDs are routinely placed immediately following placental delivery.support this hypothesis. A recent study published in 2010 by Chen et al. showed an approximately 24% expulsion rate.

Six week postpartum IUD placement for contraception will be compared to immediate post-placental IUD placement, to determine whether immediate IUD insertion after delivery has an acceptably low rate of expulsion, infection, perforation and unintended pregnancy, and a high rate of retention, patient satisfaction, and maintenance of contraception.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 15- 45 years of age and received their prenatal care at the University of Louisville OB/GYN clinic
2. Planned vaginal delivery
3. Negative third trimester cultures for Gonorrhea and Chlamydia
4. Desire to use the IUD for contraception

Exclusion Criteria:

1. Uterine anomalies
2. Uterine or cervical neoplasia
3. Past or current breast cancer
4. Chorioamnionitis
5. Acute liver disease
6. Postpartum hemorrhage lasting greater than ten minutes or more than 500 mL blood loss
7. Received prenatal other than at the University of Louisville OB/GYN Clinic
8. Cesarean section

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2009-07; Primary Completion 2011-03-21 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Stauble, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- IUD Insertion 6 Weeks After Delivery: Device:Levonorgestrel-releasing intrauterine device marketed as Mirena. Subjects randomized to interval placement will have their IUD placed in the office at six weeks postpartum or later. They must return for one visit within a month for a "string check"
- Immediate Post-Placental Insertion: Device: Levonorgestrel-releasing intrauterine device marketed as Mirena Subjects randomized to immediate post-placental placement within 10 minutes of delivery will have an IUD placed manually under sterile technique and with ultrasound guidance. An ultrasound will be performed within two days postpartum to verify proper placement and again at approximately six weeks postpartum
Period: Overall Study
Arm/Group | IUD Insertion 6 Weeks After Delivery | Immediate Post-Placental Insertion
Started | 11 | 21
Patients Who Received IUD | 0 (Subjects did not return at 6 weeks for IUD insertion.) | 18
Patients Returned for 6 wk Postpartum | 0 | 2
Completed | 0 | 0
Not Completed | 11 | 21
Not completed — Lost to Follow-up | 10 | 17
Not completed — Physician Decision | 1 | 2
Not completed — IUD expelled before month 6 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- IUD Insertion 6 Weeks After Delivery: Subjects randomized to interval placement will have their IUD placed in the office at six weeks postpartum or later.
- Immediate Post-placental Insertion: Subjects randomized to immediate post-placental placement within 10 minutes of delivery will have an IUD placed
- Total: Total of all reporting groups
Arm/Group | IUD Insertion 6 Weeks After Delivery | Immediate Post-placental Insertion | Total
Number analyzed (Participants) | 11 | 21 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 21 | 32
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 21 | 32
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 21 | 32

OUTCOME MEASURES:

1. Primary Outcome: IUD Expulsion Rate
Description: The investigators wanted to compare the expulsion rate of IUDs between the two treatment arms: immediate placement after placental delivery and interval placement 6 weeks after delivery. IUD expulsion is confirmed by the inability of the physician to visualize the string attached to the IUD coming from the cervix.
Time Frame: 6 months
Population: 0 participants were evaluable in the Arm "IUD Insertion 6 Weeks After Delivery", as 0 participants received an IUD at 6 weeks, and 2 participants in the Arm "Immediate Post-placental Insertion" were evaluable, as there were only 2 participants that came back for a follow up appointment.
Measure: Count of Participants; unit: Participants
Groups:
- IUD Insertion 6 Weeks After Delivery: Subjects randomized had their IUD placed in the office at six weeks postpartum or later.
- Immediate Post-placental Insertion: Subjects randomized to immediate post-placental placement within 10 minutes of delivery had an IUD placed manually under sterile technique and with ultrasound guidance
Arm/Group | IUD Insertion 6 Weeks After Delivery | Immediate Post-placental Insertion
Number analyzed (Participants) | 0 | 2
Participants | 0 | 2

ADVERSE EVENTS:
Arm/Group | IUD Insertion 6 Weeks After Delivery | Immediate Post-placental Insertion
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/21
Other Adverse Events (participants affected / at risk) | 0/11 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes